CLINICAL TRIAL: NCT00255944
Title: Internet-based Efficacy Trial of an HIV Prevention Program
Brief Title: Effectiveness of an Online Prevention Program in Reducing the Risk of STD Infection in Young Adults
Acronym: Youthnets
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 02-0764b; R01MH063690 (NIH); DAHBR 9A-ASI
Record Dates: First submitted 2005-11-16; First posted 2005-11-21 (Estimated); Results first posted 2020-10-05 (Actual); Last update posted 2020-10-05 (Actual); Status verified 2020-09

CONDITIONS: HIV Infections; Sexually Transmitted Diseases
Keywords: HIV Prevention; Internet Intervention; STDs
MeSH Terms: conditions — HIV Infections; Sexually Transmitted Diseases

ARMS (2):
- Youthnet messages on Facebook (Experimental): Participants will receive internet-based messages from the Youthnet program
  Interventions: Behavioral: Youthnet Internet-based program
- Messages on Facebook about current events (Active Comparator): Participants will receive internet-based messages from the control program
  Interventions: Behavioral: Control Internet based program

INTERVENTIONS:
Behavioral: Youthnet Internet-based program — Messages from the Youthnet program will be interactive and tailored specifically to HIV/STD risk reduction. Participants will be exposed to five flash computer vignettes of 30 seconds each, concerning condom attitudes, norms self-efficacy, and risk awareness.
  Arms: Youthnet messages on Facebook
Behavioral: Control Internet based program — The control program will deliver standard STD/HIV prevention messages.
  Arms: Messages on Facebook about current events

SUMMARY:
This study will evaluate the effectiveness of a tailored interactive online risk reduction program versus a standard online risk reduction program in reducing the risk of Sexually Transmitted Diseases (STD) infection in young adults.

DETAILED DESCRIPTION:
Adolescents and young adults are at the greatest risk for acquiring an STD. Approximately 3 million people between the ages of 18 and 24 become infected each year. Education about the risks and consequences of unprotected sex is a powerful tool that can be used to prevent or reduce the risk of infection. The program in this study will deliver messages to educate participants about condom use and the risk of STD infection. This study will evaluate the effectiveness of a tailored interactive online risk reduction program versus a standard online risk reduction program in reducing the risk of STD infection in young adults.

Participants in this 1-year open-label study will be recruited exclusively via the internet. Participants will be randomly assigned to receive internet-based messages from either the Youthnet program or the control program. Messages from the Youthnet program will be interactive and tailored specifically to Human Immunodeficiency Virus/Sexually Transmitted Diseases (HIV/STD) risk reduction. The control program will deliver standard STD/HIV prevention messages. Participants will be assessed at baseline and a follow-up session 4 months after enrollment. Frequency of condom use and attitudes toward condom use will be assessed using behavioral scales.

ELIGIBILITY:
Inclusion Criteria:

* Has access to the internet
* Has an e-mail address

Exclusion Criteria:

* Colorado resident

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 2622 (Actual)
Dates: Start 2005-10; Primary Completion 2008-11 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sheana Bull, PhD, Principal Investigator — University of Colorado, Denver
Locations (1):
- Internet-Based, accessible from anywhere, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Intervention Arm--exposure to Intervention on Facebook: Participants will receive internet-based messages from the Youthnet program
  Youthnet Internet-based program: Messages from the Youthnet program will be interactive and tailored specifically to HIV/STD risk reduction. Participants will be exposed to five flash computer vignettes of 30 seconds each, concerning condom attitudes, norms self-efficacy, and risk awareness.
- Control Arm--exposure to Control Content on Facebook: Participants will receive internet-based messages from the control program
  Control Internet based program: The control program will deliver standard STD/HIV prevention messages.
Period: Overall Study
Arm/Group | Intervention Arm--exposure to Intervention on Facebook | Control Arm--exposure to Control Content on Facebook
Started | 1311 | 1311
Completed | 514 | 477
Not Completed | 797 | 834
Not completed — Lost to Follow-up | 797 | 834

BASELINE CHARACTERISTICS:
Groups:
- Intervention: Participants will receive internet-based messages from the Youthnet program
  Youthnet Internet-based program: Messages from the Youthnet program will be interactive and tailored specifically to HIV/STD risk reduction. Participants will be exposed to five flash computer vignettes of 30 seconds each, concerning condom attitudes, norms self-efficacy, and risk awareness.
- Control: Participants will receive internet-based messages from the control program
  Control Internet based program: The control program will deliver standard STD/HIV prevention messages.
- Total: Total of all reporting groups
Arm/Group | Intervention | Control | Total
Number analyzed (Participants) | 514 | 477 | 991
Age, Continuous [Mean (Standard Deviation); unit: years] | 21.7 (1.8) | 21.8 (1.8) | 21.7 (1.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 230 | 234 | 464
  Male | 284 | 243 | 527
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 15 | 7 | 22
  Not Hispanic or Latino | 499 | 470 | 969
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 103 | 86 | 189
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 11 | 11 | 22
  White | 335 | 316 | 651
  More than one race | 31 | 31 | 62
  Unknown or Not Reported | 34 | 33 | 67

OUTCOME MEASURES:

1. Primary Outcome: Efficacy of Internet-based Program for Increasing Condom Use With Non-main Sex Partners
Time Frame: Month 2 post baseline
Measure: Mean (Standard Deviation); unit: percentage of sex acts protected by cond
Groups:
- Intervention Arm--exposure to Facebook: Participants will receive internet-based messages from the Youthnet program
  Youthnet Internet-based program: Messages from the Youthnet program will be interactive and tailored specifically to HIV/STD risk reduction. Participants will be exposed to five flash computer vignettes of 30 seconds each, concerning condom attitudes, norms self-efficacy, and risk awareness.
Arm/Group | Intervention Arm--exposure to Facebook | Control Arm--exposure to Control Content on Facebook
Number analyzed (Participants) | 514 | 447
percentage of sex acts protected by cond | .68 (1.96) | .56 (1.96)

2. Secondary Outcome: Efficacy of Internet-based Program for Increasing Condom Use Attitudes, Norms, and Intentions With Non-main Sex Partners
Time Frame: Month 2 post baseline
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Intervention Arm--exposure to Intervention on Facebook | Control Arm--exposure to Control Content on Facebook
Serious Adverse Events (participants affected / at risk) | 0/1311 | 0/1311
Other Adverse Events (participants affected / at risk) | 0/1311 | 0/1311

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No